CLINICAL TRIAL: NCT00232232
Title: Use of Fish Oils to Prevent Atrial Mechanical Stunning and Atrial Remodeling Due to Atrial Arrhythmia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003.074
Record Dates: First submitted 2005-10-02; First posted 2005-10-04 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial mechanical stunning and; atrial electrical remodeling
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Fish Oils

ARMS (2):
- Control (No Intervention): No fish oil
- Fish oil (Experimental): Patients prescribed 6g/day of fish oil containing 1.8g EPA+DHA in a 1.5:1 ratio
  Interventions: Drug: Fish oil

INTERVENTIONS:
Drug: Fish oil
  Arms: Fish oil

SUMMARY:
The purpose of this study is to investigate whether fish oils may be of benefit to patients with certain heart rhythm disturbances called atrial fibrillation and atrial flutter.

Atrial fibrillation and atrial flutter are two heart conditions that can be successfully treated in the hospital by an ablation (in the case of atrial flutter) or a cardioversion (in the case of atrial fibrillation). Ablation involves the application of high frequency energy waves to a particular spot in the heart. Cardioversion involves resetting the heart back to a normal rhythm with the use of an electric current.

Fish oil supplements may be of benefit to patients with heart problems. Recent evidence suggests that fish oils may benefit those with rhythm disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Chronic atrial flutter requiring radiofrequency ablation.
* Chronic atrial fibrillation requiring internal cardioversion.

Exclusion Criteria:

* Sinus rhythm.
* Pregnancy.
* Patients > 80 years and < 18 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-09; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The extent of left atrial stunning in fish oil group compared to control after reversion of atrial arrhythmias to sinus rhythm. | 18 months

OTHER OUTCOMES:
Adverse events related to fish oil ingestion. | 18 months
  Tolerability, mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sparks, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Kumar S, Sutherland F, Wheeler M, Heck PM, Lee G, Teh AW, Garg ML, Morgan JG, Sparks PB. Effects of chronic omega-3 polyunsaturated fatty acid supplementation on human atrial mechanical function after reversion of atrial arrhythmias to sinus rhythm: reversal of tachycardia-mediated atrial cardiomyopathy with fish oils. Heart Rhythm. 2011 May;8(5):643-9. doi: 10.1016/j.hrthm.2011.01.014. Epub 2011 Jan 11. PMID 21232631